CLINICAL TRIAL: NCT01075737
Title: Observational Study to Assess the Quality of Life of the Caregivers of Patients With Multiple Sclerosis
Brief Title: An Observational Study to Assess the Quality of Life of the Patients With Multiple Sclerosis and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 200077-501
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Sclerosis; Quality of life
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with Multiple Sclerosis: Subjects with diagnosed MS according to the revised Mc Donald criteria 2005; aged >21 years.
- Caregivers: Caregivers (aged >21 years) for MS subjects.

SUMMARY:
This is an observational, non controlled, non-interventional, multicentric, prospective study planned to be conducted in 450 subjects diagnosed with MS and their caregivers in 20 centres of Argentina. The observations from this study will contribute to the awareness of the impact on the Quality of Life (QoL) of the caregivers and, eventually will also provide measures for helping the subjects with multiple sclerosis (MS) without leaving aside the care of the physical and psychic health of those who work as caregivers.

DETAILED DESCRIPTION:
Caregivers of subjects diagnosed with MS have to take care of many activities of MS subjects that they cannot perform themselves, because of their lack of autonomy. The fact of aiding a person with some degree of disability due to a chronic disease in an intense way and for a long time could generate a high level of satisfaction in the caregiver; but at the same time the emotional and physical exhaustion of the caregiver increases as the disease progresses. The QoL of the person who is emotionally bonded to the MS subject as a caregiver has a great chance to be affected; and this is for sure more likely than in the case when the caregiver is a hired professional.

OBJECTIVES

Primary objective:

* To identify the impact of MS on the QoL of the MS subjects and their caregivers

Secondary objectives:

* To establish the correlation between the QoL of the subjects with MS and their caregivers
* To identify the predictors of the QoL in the caregiver group

This is an observational, prospective and non-interventional study planned to be conducted in 20 centers in Argentina. The subjects with diagnosed MS will be managed with the clinical and therapeutic elements that their treating doctors considered appropriate, without modifying their decisions due to the subjects' inclusion into the study. The caregivers will be asked to complete the QoL questionnaire as a part of the normal interview on each and every visit. The total duration of the study is 24 months. A descriptive analysis will be performed for the demographic and clinical characteristics of the investigation subjects, as well as for the characteristics of the treatments they receive when they start their participation in this study. For the qualitative variables, treatment modifications, frequency tables and the percentages will be performed.

ELIGIBILITY:
Inclusion Criteria:

* MS subjects and their caregivers, >21 years of age of both sexes
* Subjects who have signed informed consent
* Subjects with established MS diagnosis according to the revised Mc Donald criteria - 2005 with at least 1 year of evolution
* Subjects with MS that have an identified caregiver

Exclusion Criteria:

* Subjects with other(s) associated neurological, psychiatric or systemic disease(s)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with diagnosed MS and their caregivers in Argentinean population.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Impact of MS on QoL of subjects diagnosed with multiple sclerosis (MS) and their caregivers | Each visit starting from the initial visit (Day 0) to end of the observation period (i.e. 24 months)
  SF-36 will be administered to subjects diagnosed with MS and their caregivers; Beck depression inventory and MS-Functional system scores to subjects diagnosed with MS.

SECONDARY OUTCOMES:
Correlation between QoL of subjects with MS and their caregivers | During the observation period of 24 months starting from the initial visit (i.e. Day 0)
Predictors of QoL of caregivers | During the observation period of 24 months starting from the initial visit (i.e. Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Jacobo, Neurologist, Principal Investigator — 25 de Mayo 138 (Capital, Pcia. de Santiago del Estero) G4200AWD
Locations (1):
- 25 de Mayo 138, Capital, Pcia. de, Santiago del Estero, Argentina